CLINICAL TRIAL: NCT00000118
Title: Ganciclovir Implant Study for Cytomegalovirus Retinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-14
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome; Cytomegalovirus Retinitis
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Cytomegalovirus Retinitis

INTERVENTIONS:
Device: Sustained-Release Intraocular Drug Delivery System

SUMMARY:
To determine the therapeutic efficacy of a sustained-release intraocular drug delivery system for ganciclovir therapy of cytomegalovirus (CMV) retinitis in patients with acquired immunodeficiency syndrome (AIDS).

DETAILED DESCRIPTION:
CMV retinitis occurs in 20 to 30 percent of patients with AIDS and is the leading cause of visual loss in these patients. At present, ganciclovir and foscarnet are the only drugs that have been approved by the U.S. Food and Drug Administration for the treatment of CMV retinitis. The therapeutic regimen for each drug consists of a 2-week induction period followed by daily maintenance intravenous infusions. Unfortunately, CMV retinitis usually progresses despite daily maintenance therapy, and both drugs are associated with significant systemic toxicity that often limits their therapeutic usefulness. As an alternative to intravenous administration, direct intravitreal injections of ganciclovir have been studied and have been shown to be effective in delaying the progression of CMV retinitis. The short half-life of the drug, however, necessitates one to two intraocular injections a week to maintain therapeutic levels. Widespread adoption of this technique has been limited because of the logistical difficulties and inherent risks associated with numerous intravitreal injections.

A drug delivery system capable of continuous delivery of ganciclovir into the vitreous cavity has been developed. The device consists of a 6-mg pellet of ganciclovir that is coated with a series of polymers with variable permeability to ganciclovir. The device is surgically implanted through the pars plana.

Thirty eyes of 26 patients with unilateral non-sight-threatening CMV retinitis were randomly assigned to one of two groups: (1) immediate therapy with a device designed to release ganciclovir into the vitreous cavity a over approximately a 4-month period or (2) deferred treatment. In patients with bilateral non-sight-threatening CMV retinitis, one eye was randomly assigned to receive a ganciclovir implant with the other eye assigned to deferred treatment. (Note: The original trial design included a third randomized arm using a 2 ug/hour device. This arm was dropped for logistical reasons after enrolling two patients.)

Patients assigned to immediate treatment underwent surgery to implant the ganciclovir device within 48 hours of enrollment and baseline photographs. Postoperatively, patients were evaluated the next day, weekly for 2 weeks, and then every 2 weeks until progression of CMV retinitis occurred. At each examination, in both eyes, visual acuity with current correction and best correction was determined using Early Treatment Diabetic Retinopathy Study eye charts; intraocular pressure was determined; evidence of inflammation or cataract was evaluated; and all retinal findings were documented. Any adverse event considered even possibly related to the device or to the implantation procedure was documented. Standardized nine-field fundus photographs were taken at each 2-week visit. The ganciclovir implant was exchanged at 32 weeks or earlier if progression of CMV retinitis occurred.

The primary end point was time to CMV retinitis progression, defined as the time (days) from initiating therapy until the advancement of 750-um over a 750 um front of any border of any lesion was observed. Standardized nine-field photographs were taken at 2-week intervals and analyzed in a masked fashion by the Fundus Photograph Reading Center to determine evidence of CMV retinitis progression.

Secondary end points included time to development of CMV retinitis in the contralateral eye, time to development of visceral CMV, and time to death.

ELIGIBILITY:
All patients must have had AIDS as defined by the Centers for Disease Control and Prevention and non-sight-threatening CMV retinitis Patients could not have been previously treated with systemic ganciclovir or foscarnet and must not have had evidence of other organ involvement with CMV. Patients must have had an absolute neutrophil count (ANC) greater than 1,000 cells/mL and a platelet count greater than 25,000/mm3

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-10; Study Completion 1993-12 (Actual)

REFERENCES:
- [Background] Martin DF, Parks DJ, Mellow SD, Ferris FL, Walton RC, Remaley NA, Chew EY, Ashton P, Davis MD, Nussenblatt RB. Treatment of cytomegalovirus retinitis with an intraocular sustained-release ganciclovir implant. A randomized controlled clinical trial. Arch Ophthalmol. 1994 Dec;112(12):1531-9. doi: 10.1001/archopht.1994.01090240037023. PMID 7993207